CLINICAL TRIAL: NCT05138354
Title: Standard Care Combined With Low-Level Laser Therapy and Myofascial Release Versus Standard Care Alone in Pregnant Women With Temporomandibular Disorder: A Randomized Controlled Trial
Brief Title: Standard Care With LLLT & Myofascial Release Versus Standard Care Alone in Pregnant Women With Temporomandibular Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTMD2021
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy; Myofascial Release Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients received a 4-week treatment program (12 treatment sessions, three times a week). Patients received the conservative treatment protocol comprised of ultrasound, hot pack application, and exercises.
  Interventions: Other: Standard care
- Intervention group (Experimental): Patients received a 4-week treatment program (12 treatment sessions, three times a week). Patients received LLLT and myofascial release combined with the control intervention. the conservative treatment protocol comprised of ultrasound, hot pack application, and exercises
  Interventions: Other: Low Level laser therapy; Other: Myofascial release; Other: Standard care

INTERVENTIONS:
Other: Low Level laser therapy — MLS® device (ASA Srl, Vicenza, Italy) IR laser with two synchronized sources (laser diodes) and a wavelength of 808 nm to deliver the intervention. The laser probe will be held vertically in contact with the skin to deliver the irradiation at three mandibular condyle points (front, behind and over) and one point at the external acoustic meatus. The irradiation will be applied with a laser bean of 3.14 cm² diameter for 14 seconds at each place using a pulse rate of 1500 Hz, pulse duration of 100ns, and energy density: 16 J/cm².
  Arms: Intervention group
Other: Myofascial release — Patients will be positioned in supine in a treatment table. The therapist seated beside the patient at the side of affected temporomandibular joint to apply gross release technique for masseter, pterygoid and temporalis muscles. At each point, the therapist applied the technique for 90 seconds and repeated 5 times during the session (5 seconds of rest between each repetition).(15) The therapist worn gloves to deliver the intraoral myofascial release. In case the patient reported any latex allergies, the gloves were replaced by a latex free model.
  Arms: Intervention group
Other: Standard care — 1. Ultrasound Participants will receive an application of pulsed ultrasound at a frequency of 3 MHz and an intensity of 0.5 W/cm² with a 1:1 duty cycle over TMJ for six minutes.
  2. Hot pack Participants will receive a warm water pack the TMJ and masticatory muscles for 10 minutes.
  3. Exercise program:
  Active exercises for mandibular muscles will be used to correct the mouth opening
  1. Lateral movements of the jaw (3 sets of 10 repetitions).
  2. Jaw relaxation exercise (3 sets of 10 repetitions).
  3. Chin tuck (10 repetitions, holding 10s each).
  4. Resisted opening of the mouth (3 sets of 10 repetitions).
  5. Resisted closing of the mouth (3 sets of 10 repetitions).
  6. Stretching exercise for mandibular muscles.

SUMMARY:
This study will investigate a novel approach to treat pregnant women with tempromandibular disorder using a combined method of low level laser therapy, myofascial release and standard care versus standard care alone. It's hopeful that the results of this study can fill the gap of knowledge surrounding the conservative treatment options for TMD in order to help patients restore their oral function properly and promote new ways of addressing TMD.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with myofascial TMD according to the Research Diagnostic Criteria for Temporomandibular Disorders

Exclusion Criteria:

* facial neuro-musculoskeletal pathologies (i.e., facial trauma and/or fractures, and bell's palsy)
* acute infections or systemic disorders
* osteoporosis
* cervical spine or upper limb dysfunction
* steroid infiltration4
* any recent dental treatment taken or surgery over TMJ
* hypermobile joint
* neurological impairments

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Changes in visual analogue scale | Baseline and after 4 weeks
  Visual analog scale (VAS), a grading scale range from 0 to 100 mm. 0 mm represented no pain or discomfort at all and 100 mm represented the greatest amount of pain or discomfort imaginable. Participant drew a line that intersects the grading scale to show the amount of pain or discomfort that he or she experienced at that moment. The assessor then used a ruler to measure the length from 0 mm to the intersecting line and recorded the value.
Changes in pain pressure threshold (PPT) | Baseline and after 4 weeks
  Comparing pain pressure threshold differences on both sides over TMJ, masseter and anterior temporalis.

SECONDARY OUTCOMES:
Limitations of daily function in temporomandibular disorder questionnaire | Baseline and after 4 weeks
  The limitations in daily functions in the temporomandibular disorder questionnaire (LDF-TMDQ) assess participants' functionality by asking them to report how much the jaw problem prevents or limits their performance in a list of 10 daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Radwa M Yehia, Ph.D, Study Director — Faculty of Physical Therapy, October 6 University
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trial and after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 Months after study publication
Access Criteria: Email: mohamed.magdy.pt@o6u.edu.eg